CLINICAL TRIAL: NCT05658926
Title: A Brief Intervention for Patients on Opioids for Acute Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Lisa Matero, Senior Staff Psychologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS Acute Pain
Record Dates: First submitted 2017-07-31; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Mindfulness; Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will learn a brief, mindfulness skill
  Interventions: Behavioral: Mindfulness
- Education (Placebo Comparator): Participants will receive education about the effects of emotions on pain
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Mindfulness — Patients will learn how to use diaphragmatic breathing with mindfulness
  Arms: Intervention
Other: Education — Patients will be provided with education regarding the Gate Control Theory of Pain.
  Arms: Education

SUMMARY:
This study aims to evaluate benefits of a brief intervention for patients who are prescribed opioids for acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to Henry Ford Hospital
* Patients who have been evaluated by the Psychosomatic Medicine Service
* Patients who are prescribed at least one opioid for an acute pain condition

Exclusion Criteria:

* Patients taking an opioid for a chronic pain condition within the previous year
* History of an opioid use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Pain severity | Change from pre- to post-intervention. The intervention is approximately 10 minutes so the measurements are taken about 10 minutes apart.
  Pain severity rated on a 0-10 scale

SECONDARY OUTCOMES:
Stress level | Change from pre- to post-intervention. The intervention is approximately 10 minutes so the measurements are taken about 10 minutes apart
  Stress level rated on a 0-10 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States